CLINICAL TRIAL: NCT01869491
Title: A Multi-centre, Randomised, Double-blind, Two Arm, Parallel Group, Placebo-controlled Study to Assess the Effect of Compound Sodium Alginate Double Action Chewable Tablets in Patients With Gastro-esophageal Reflux Disease
Brief Title: Compound Sodium Alginate Double Action Chewable Tablet Symptomatic Relief Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA1210
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2025-03-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Gastroesophageal Reflux Disease; Dyspepsia
Keywords: Gastroesophageal Reflux Disease; GERD; Dyspepsia; Indigestion; Heartburn; Acid reflux; Compound Sodium Alginate Double Action Chewable Tablets; Gaviscon Double Action Tablets
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia; Heartburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Alginate Double Action Chewable Tablets (Active Comparator): Compound Sodium Alginate Double Action Chewable Tablets, 2 tablets four times daily
  Interventions: Drug: Compound Sodium Alginate Double Action Chewable Tablets
- Matching placebo tablets (Placebo Comparator): Matching placebo tablets, 2 tablets four times daily
  Interventions: Drug: Matching placebo tablets

INTERVENTIONS:
Drug: Compound Sodium Alginate Double Action Chewable Tablets — 2 tablets four times daily
  Other Names: Gaviscon Double Action Tablets
  Arms: Sodium Alginate Double Action Chewable Tablets
Drug: Matching placebo tablets — 2 tablets four times daily
  Other Names: Placebo
  Arms: Matching placebo tablets

SUMMARY:
This study is being conducted to provide evidence that Compound Sodium Alginate Double Action Chewable Tablets are effective in managing the symptoms of heartburn, acid regurgitation and dyspepsia in patients with Gastroesophageal Reflux Disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* Current evidence of symptomatic GERD in accord with the Montreal definition.
* Patients must have had troublesome heartburn and/or regurgitation (with or without dyspepsia symptoms) of at least mild or moderate intensity on at least 5 days during the week before the start of screening.

Exclusion Criteria:

* Patients who have a history of drug, solvent or alcohol abuse.
* Patients who have suffered cardiac chest pain within the last year.
* Patients who have suffered a recent, significant unexplained weight loss of more than 6 kg in the last 6 months.
* Female patients of childbearing potential who, for the duration of the study, are either unwilling or unable to take adequate contraceptive precautions or are unwilling to be sexually abstinent.
* Pregnancy or lactating mother.
* Patients with a history and/or symptom profile suggestive of the following: any other gastrointestinal (GI) disease, erosive GERD (Los Angeles classification grades C-D), Barrett's oesophagus, acute peptic ulcer and/or ulcer complications, Zollinger-Ellison syndrome, gastric carcinoma, pyloric stenosis, oesophageal or gastric surgery, intestinal obstruction, current pernicious anaemia, indication for H. pylori eradication therapy, known gastrointestinal bleeding (hematochezia or hematemesis) within 3 months prior to the study, and severe diseases of other major body systems.
* Patients who were observed at screening to have a hiatus hernia with a diameter which exceeds 3 cm.
* Patients who have taken anti-cholinesterase drugs, traditional Chinese medicines for treating gastrointestinal disease, ulcermin or misoprostol preparations within 7 days prior to screening or throughout the study.
* Patients who have taken proton pump inhibitors (PPIs) during the 10 days prior to screening, prokinetics or H2 antagonists during the 5 days prior to screening or systemic glucocorticosteroids, non-steroidal anti-inflammatory drugs (except for low dose aspirin which can be given for cardioprotection) on more than 3 consecutive days or PPI-based triple or quadruple therapy for eradication of H-pylori during the last 28 days.
* Patients taking or requiring to take macrolide antibiotics, such as erythromycin, azithromycin, from the day before screening.
* Patients with known hypophosphataemia, phenylketonuria or hypercalcaemia.
* Patients with severe constipation, or history of intestinal obstruction.
* In the opinion of the Investigator, patients with damaged heart or kidney function and patients who require a low sodium diet.
* Any previous history of allergy or known intolerance to any of the investigational medicinal products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1107 (Actual)
Dates: Start 2013-06-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yaozong, MD, PhD, Principal Investigator — Shanghai Jiao Tong University, School of Medicine, Shanghai, China
Locations (2):
- China (2):
  - RB Investigational Sites, Beijing
  - RB Investigational Sites, Shanghai

REFERENCES:
- [Derived] Sun J, Yang C, Zhao H, Zheng P, Wilkinson J, Ng B, Yuan Y. Randomised clinical trial: the clinical efficacy and safety of an alginate-antacid (Gaviscon Double Action) versus placebo, for decreasing upper gastrointestinal symptoms in symptomatic gastroesophageal reflux disease (GERD) in China. Aliment Pharmacol Ther. 2015 Oct;42(7):845-54. doi: 10.1111/apt.13334. Epub 2015 Jul 31. PMID 26228097 (Retraction: PMID 30318684 Aliment Pharmacol Ther. 2018 Nov;48(9):1039)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Started | 552 | 555
Completed | 531 | 531
Not Completed | 21 | 24
Not completed — Adverse Event | 3 | 5
Not completed — Lack of Efficacy | 0 | 3
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Lost to Follow-up | 11 | 9
Not completed — No further need of investigational product | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eight subjects (3 in the Sodium Alginate Double Action Chewable Tablets group and 5 in the matching placebo tablets group) were randomized in the study, but not treated, and therefore not included in the safety population, from which baseline data were drawn.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets | Total
Number analyzed (Participants) | 549 | 550 | 1099
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (11.81) | 44.8 (11.84) | 44.9 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 262 | 542
  Male | 269 | 288 | 557
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 0 | 1
  Asian | 548 | 550 | 1098
  Afro-Caribbean | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 549 | 550 | 1099

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Reflux Disease Questionnaire (RDQ) Scores for the GERD Dimension
Description: The primary study endpoint is the change from baseline in RDQ symptom scores for the GERD dimension (heartburn and regurgitation) after a 7-day treatment period of Compound Sodium Alginate Double Action Chewable Tablets compared with a matched placebo. The RDQ is a 12-item self-administered questionnaire designed to assess the frequency and severity of heartburn, acid regurgitation and dyspepsia symptoms, with a minimum score of 0 and a maximum score of 60, with lower RDQ scores showing an improved outcome. The heartburn and acid regurgitation subscales can be combined into a GERD dimension, which has a minimum score of 0 and a maximum score of 40, with lower RDQ scores showing an improved outcome.
Time Frame: 7 days
Population: Data are from patients in the intent-to-treat population, which included all patients who were recruited into the study and had at least partially completed RDQ questionnaire for the trial therapy period or were known to have withdrawn from the study due to poor efficacy.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 536 | 537
score on a scale | -1.27 [-1.37 to -1.16] | -1.06 [-1.17 to -0.95]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.31 to -0.11]

2. Secondary Outcome: Change From Baseline in RDQ Scores for the Dyspepsia Dimension
Description: The change from baseline in RDQ symptom scores for the dyspepsia dimension after a 7-day treatment period of Compound Sodium Alginate Double Action Chewable Tablets compared with a matched placebo. The dyspepsia subscale of the RDQ has a minimum score of 0 and a maximum score of 20, with lower RDQ scores showing an improved outcome.
Time Frame: 7 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 536 | 537
score on a scale | -0.98 [-1.10 to -0.86] | -0.80 [-0.91 to -0.68]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.29 to -0.08]

3. Secondary Outcome: Change From Baseline in RDQ Scores for the Heartburn Dimension
Description: The change from baseline in RDQ symptom scores for the heartburn dimension after a 7-day treatment period of Compound Sodium Alginate Double Action Chewable Tablets compared with a matched placebo. The heartburn subscale of the RDQ has a minimum score of 0 and a maximum score of 20, with lower RDQ scores showing an improved outcome.
Time Frame: 7 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 536 | 537
score on a scale | -1.16 [-1.28 to -1.04] | -0.95 [-1.07 to -0.83]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.32 to -0.10]

4. Secondary Outcome: Change From Baseline in RDQ Scores for the Regurgitation Dimension
Description: The change from baseline in RDQ symptom scores for the regurgitation dimension after a 7-day treatment period of Compound Sodium Alginate Double Action Chewable Tablets compared with a matched placebo. The regurgitation subscale of the RDQ has a minimum score of 0 and a maximum score of 20, with lower RDQ scores showing an improved outcome.
Time Frame: 7 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 536 | 537
score on a scale | -1.37 [-1.48 to -1.26] | -1.16 [-1.27 to -1.05]
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.32 to -0.09]

5. Secondary Outcome: Overall Treatment Evaluation (OTE) as a Measure of Patient Responsiveness/Satisfaction: Question 1 - Patient's Evaluation of the Change in Symptoms Over the Last 7 Days
Description: Comparison between the 2 cohorts (Compound Sodium Alginate Double Action Chewable Tablets and matching placebo) in OTE as a measure for patient's responsiveness/satisfaction, determined at Visit 3, the end-of-study visit.
  Question 1 of the OTE assessed how the patients rated their responsiveness/satisfaction on a 15-point scale (from -7 = a very great deal worse to +7 = a very great deal better).
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 536 | 537
Participants
  -7 = A very great deal worse | 0 | 0
  -6 = A great deal worse | 0 | 1
  -5 = A good deal worse | 0 | 0
  -4 = Moderately worse | 0 | 3
  -3 = Somewhat worse | 6 | 2
  -2 = A little worse | 3 | 10
  -1 = Almost the same, hardly any worse at all | 2 | 4
  0 = No change | 41 | 64
  1 = Almost the same, hardly any better at all | 32 | 47
  2 = A little better | 85 | 106
  3 = Somewhat better | 87 | 89
  4 = Moderately better | 88 | 72
  5 = A good deal better | 116 | 92
  6 = A great deal better | 53 | 33
  7 = A very great deal better | 23 | 13
  Missing | 0 | 1
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: OTE as a Measure of Patient Responsiveness/Satisfaction: Question 2 - Patient's Evaluation of the Importance of the Change in Symptoms
Description: Comparison between the 2 cohorts (Compound Sodium Alginate Double Action Chewable Tablets and matching placebo) in OTE as a measure for patient's responsiveness/satisfaction, determined at Visit 3, the end-of-study visit.
  Question 2 of the OTE addressed how patients perceived the importance of the change of the clinical status on a 7-point scale (from 1 = not important to 7 = extremely important).
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 536 | 537
Participants
  1 = Not important | 19 | 25
  2 = Slightly important | 31 | 51
  3 = Somewhat important | 48 | 44
  4 = Moderately important | 55 | 49
  5 = Important | 174 | 153
  6 = Very important | 138 | 118
  7 = Extremely important | 31 | 32
  Missing | 40 | 65
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p = 0.0433, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: For Patients With Improvement Only: OTE as a Measure of Patient Responsiveness/Satisfaction: Question 2 - Patient's Evaluation of the Importance of the Change in Symptoms
Description: For patients with improvement only, comparison between the 2 cohorts (Compound Sodium Alginate Double Action Chewable Tablets and matching placebo) in OTE as a measure for patient's responsiveness/satisfaction, determined at Visit 3, the end-of-study visit.
  Question 2 of the OTE addressed how patients perceived the importance of the change of the clinical status on a 7-point scale (from 1 = not important to 7 = extremely important).
Time Frame: 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
Number analyzed (Participants) | 484 | 452
Participants
  1 = Not important | 18 | 22
  2 = Slightly important | 29 | 48
  3 = Somewhat important | 47 | 40
  4 = Moderately important | 55 | 49
  5 = Important | 169 | 151
  6 = Very important | 136 | 112
  7 = Extremely important | 30 | 30
Statistical Analysis 1: Comparison: Sodium Alginate Double Action Chewable Tablets vs Matching Placebo Tablets; Test type: Superiority; p = 0.0503, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 8 days, from after the first dose of IMP until no later than the day of the last dose of IMP +1
Arm/Group | Sodium Alginate Double Action Chewable Tablets | Matching Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/549 | 0/550
Serious Adverse Events (participants affected / at risk) | 1/549 | 0/550
Other Adverse Events (participants affected / at risk) | 0/549 | 0/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Alginate Double Action Chewable Tablets (N=549) | Matching Placebo Tablets (N=550)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT01869491/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT01869491/SAP_001.pdf